CLINICAL TRIAL: NCT05513170
Title: Graftless Closed Sinus Tenting Using Dental Implants After Densah Burs Osteotomy Versus Conventional Osteotomy in Localized Sinus Pneumatization: a Randomized Clinical Trial
Brief Title: Closed Sinus Tenting Using Densah Burs Osteotomy Versus Conventional Osteotomy in Localized Pneumatization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Basma Mohamed Abdelfatah Mohamed Shaheen, Doctor of Dental Surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Densah Burs
Record Dates: First submitted 2022-06-27; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Edentulous Alveolar Ridge
Keywords: Densah Burs; Osteotomes; Sinus Tenting; Graftless

STUDY DESIGN:
Intervention Model Description: Patients' data will be enrolled in database of the Outpatient clinics of the Department of Oral and maxillofacial surgery, Faculty of Dentistry, Cairo University. If there is a potential eligibility, the patient will be examined thoroughly as described before. Consecutive sampling is done through screening of patients. This will continue until the target population is achieved. Identifying and recruiting potential subjects is achieved through patient database.
Who Masked: Participant, Outcomes Assessor
Masking Description: This trial is considered a randomized double blind clinical trial due to the following:
  1. The participant will be blinded to the technique that will be used during the surgical operation.
  2. The outcome assessor will be blinded
  3. The operator (DR.B.S.) will not be blinded for both techniques during the surgical operation, as the two techniques are different. (Dr. M.O.).
  The purpose of double blinding procedure is to reduce assessment bias and to increase accuracy and objectivity of clinical outcomes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed sinus lift using Densah bur (Active Comparator): Closed sinus lifting will be performed using densah burs and then dental implants will be placed.
  Interventions: Procedure: Closed sinus lift using osteotomes
- Conventional closed sinus lift using osteotomes (Active Comparator): Sinus lifting will be performed using osteotomes and then dental implants will be placed.
  Interventions: Procedure: Use of Densah Burs in closed sinus lift

INTERVENTIONS:
Procedure: Use of Densah Burs in closed sinus lift — Closed sinus will be performed using Densah Burs. Densah Burs enhance bone quality through osseodensification; a process through which bone is compacted and auto-graphted in the marrow spaces and apically to elevate the sinus floor and enhance bone density.
  Arms: Conventional closed sinus lift using osteotomes
Procedure: Closed sinus lift using osteotomes — Closed sinus lift will be performed using osteotomes. Osteotomes elevate the sinus floor and enhance the bone quality.
  Arms: Closed sinus lift using Densah bur

SUMMARY:
Isolated sinus pneumatization after single tooth extraction indicate sinus lifting for proper implant placement. The conventional way of using osteotomes to elevate the sinus is annoying to patient and also does not give the needed amount of bone around the implant. Introducing new intervention of Densah Burs helps increase bone gain around implant and decrease the patient discomfort.

DETAILED DESCRIPTION:
The rehabilitation of the edentulous posterior maxilla using osseointegrated implants is often challenging due alveolar bone resorption, low bone density and maxillary sinus pneumatization. Maxillary sinus lift is one of the most common surgical techniques used for increasing the available bone volume to place implants and restore function and esthetics. Trans-crestal approach can be successfully adopted when residual bone height is at least 5 mm. Osteotome sinus floor elevation was first in 1994, and proved to be less invasive, more conservative, less time consuming, and reduces postoperative discomfort to the patient. Moreover, this technique was found to yield predictable results with success rates of at least 95%.

Osseodensification is a new surgical technique of biomechanical bone preparation performed for dental implant placement where bone is compacted and auto grafted into open marrow spaces and osteotomy site walls in outwardly expanding directions. It was reported that osseodensification increases the bone-implant contact, bone density, and primary stability. Moreover, the insertion torque peak is directly related to implant primary stability and host bone density. Furthermore, for every 9.8 N cm of torque increased, a reduction in failure rate of 20% in single-tooth implant restoration was observed.

The objective of this study is to evaluate crestal sinus elevation using osseodensification versus osteotomy clinically and radiographically in terms of marginal bone loss, primary and secondary stability and bone gain around the implant.

ELIGIBILITY:
Inclusion Criteria:

* No inflamed sinus
* Minimum alveolar ridge height 5-6 mm
* Medical free
* Both genders males and females.

Exclusion Criteria:

* Remaining alveolar ridge height is less than 5mm
* Patients should not have taken drugs, especially bisphosphonates or drugs altering bone metabolism, within 2 months before the inclusion in the study.

  * Subjected to irradiation in the head and neck area less than 1 year before implantation.
  * Patients having history of allergy to any drugs.
  * Patients who have a history of any concomitant from a major known medical problem and/or ongoing pharmacologic treatments
  * Untreated periodontitis.
  * Poor oral hygiene and motivation.
  * Uncontrolled diabetes.
  * Pregnant or nursing.
  * Substance abuse.
  * Psychiatric problems or unrealistic expectations.
  * Severe bruxism or clenching.
  * Immunosuppressed or immunocompromised.
  * Treated or under treatment with intravenous amino-bisphosphonates.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of Bone Change in Cone Beam CT | three and six months
  The amount of bone change will be determined by superimposing pre-operative CBCT (cone-beam computed tomography), three months post-operative, and six months post-operative CBCT.

SECONDARY OUTCOMES:
Measurement of Primary and Secondary Implant stability using Resonance Frequency Analysis (RFA) | At the day of implant placement and after six months
  The implant stability quotient (ISQ) of the implants will be measured using a resonance frequency analysis measuring device, that is, Ostell, at the time of placement, which is the primary stability, and after six months, which is the secondary stability. The implant stability quotient has a scale ranging from 0 to 100 in which 0 is a failed implant and 100 is maximum implant stability.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ottoni JM, Oliveira ZF, Mansini R, Cabral AM. Correlation between placement torque and survival of single-tooth implants. Int J Oral Maxillofac Implants. 2005 Sep-Oct;20(5):769-76. PMID 16274152
- [Background] Summers RB. A new concept in maxillary implant surgery: the osteotome technique. Compendium. 1994 Feb;15(2):152, 154-6, 158 passim; quiz 162. PMID 8055503
- See also: Clinical and radiographic evaluation of osseodensification versus osteotome for sinus floor elevation in partially atrophic maxilla: A prospective long term study — https://edj.journals.ekb.eg/article_71261_ed987b0840ffacb78fc722592cb620ed.pdf
- See also: Primary Stability of Implant in Closed Sinus Lifting Cases Using Densah Bur Versus Osteotome — https://clinicaltrials.gov/ct2/show/NCT03559777
- See also: Patient Perception and Radiographic Assessment of Sinus Lifting Procedure using Densah Bur versus Osteotome-mediated sinus lifting: A Randomized Clinical Trial — https://adjc.journals.ekb.eg/article_165194_0f7e7df22Scb83b2ace99f7d370d885c.pdf

DOCUMENTS (3):
  • Study Protocol (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT05513170/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT05513170/SAP_001.pdf
  • Informed Consent Form (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT05513170/ICF_002.pdf